CLINICAL TRIAL: NCT04851262
Title: Home-based Progressive Resistance Exercise to Enhance Physical Performance of Older Adults With Possible Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW20-868
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is a 12-week home-based resistance training programme with phased progression. The intervention will have three phases: (i) an initial phase focused on training the target muscle(s)/movements with minimal or no external weight; (ii) an intermediate phase targeting muscle strength with increased practice resistance; and (iii) an advanced phase targeting the further enhancement of muscle strength by challenging multiple muscle groups. Each phase will involve exercises targeting the trunk, back, hip, upper-limb and lower-limb muscles.
  Interventions: Behavioral: Exercise
- Waitlist control (Other): The waitlist control participants will start the intervention 12 weeks after the baseline assessment.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The intervention is to be taught by fitness trainer at the participants' home at the start of each phase. The exercise progression model for older adults recommended by the American College of Sports Medicine, which emphasise gradual increments in training load and systematically alter one or more programme components, will be adopted.

SUMMARY:
The overall aim of the proposed project is to improve muscle strength in older adults with possible sarcopenia by promoting home-based progressive resistance exercise. The target population for health talks is community-dwelling older adults. A Three monthly home-visits and weekly phone calls will be made. A waitlist randomised controlled trial will be conducted to evaluate effectiveness, and qualitative feedback will be collected from participants. A pilot study will be conducted first.

ELIGIBILITY:
The inclusion criteria are:

* Aged 65-89;
* Possible sarcopenia (defined by AWGS 2019);
* No cognitive impairment (Abbreviated Mental Test score ≥8); and
* No communication problems.

The exclusion criteria are:

* having engaged in a structured exercise programme in the past 6 months or planning to do so within the intervention period;
* mobility-limiting injury of the hands or lower limbs, surgery or hospitalisation within the intervention period;
* contraindications such as musculoskeletal/cardiorespiratory disorders, or any advanced diseases that inhibit them from exercising.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Change in lower-limb muscle strength at 12 weeks from baseline | 12 weeks after baseline
  Measured by Short Physical Performance Battery (SPPB), higher score indicates better performance

SECONDARY OUTCOMES:
Change in lower-limb muscle strength at 24 weeks from baseline | 24 weeks after baseline
  Measured by Short Physical Performance Battery (SPPB), higher score indicates better performance

OTHER OUTCOMES:
Change in handgrip strength at 12 weeks from baseline | 12 weeks after baseline
  Measured by a spring-type dynamometer, higher value indicates better performance
Change in handgrip strength at 24 weeks from baseline | 24 weeks after baseline
  Measured by a spring-type dynamometer, higher value indicates better performance
Status of possible sarcopenia at 12 weeks from baseline | 12 weeks after baseline
  Indicated by 5-time chair stand test ≥12 second, or men and women with <28 kg and <18 kg strength
Status of possible sarcopenia at 24 weeks from baseline | 24 weeks after baseline
  Indicated by 5-time chair stand test ≥12 second, or men and women with <28 kg and <18 kg strength
Sarcopenia risk score at 12 weeks from baseline | 12 weeks after baseline
  Measured by SARC-CalF, which is a combination of SARC-F questionnaire and calf circumference, a cut of of >=11 indicates high risk
Sarcopenia risk score at 24weeks from baseline | 24 weeks after baseline
  Measured by SARC-CalF, which is a combination of SARC-F questionnaire and calf circumference, a cut of of >=11 indicates high risk

CONTACTS AND LOCATIONS:
Locations (1):
- Community, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
To protect confidentiality of participants.